CLINICAL TRIAL: NCT00154804
Title: A Phase II Study of Concurrent Chemoradiotherapy With Twice Weekly Paclitaxel and Cisplatin (Twice Weekly TP) Followed by Surgery for Locally Advanced Esophageal Cancer
Brief Title: CCRT With Twice Weekly Paclitaxel and Cisplatin Followed by Surgery for Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 900603
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2004-04

CONDITIONS: Esophageal Cancer
Keywords: Concurrent Chemoradiotherapy; Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Paclitaxel, Cisplatin,Surgery, CCRT

INTERVENTIONS:
Drug: Paclitaxel, Cisplatin,Surgery, CCRT

SUMMARY:
CCRT with twice weekly paclitaxel and cisplatin in patient with locally advanced esophageal cancer.

DETAILED DESCRIPTION:
The purpose of this study is to find out the clinical and pathological response rates of pre-operative concurrent chemoradiotherapy (CCRT) with twice weekly paclitaxel and cisplatin in patient with locally advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven SCC or adenocarcinoma of esophagus .
2. Locally advanced esophageal cancer , defined as T3 and/or N1 disease.( AJCC 1998)
3. M1a disease defined ( AJCC 1998) , including celiac lymph node for lower thoracic esophageal cancer and cervical lymph node involvement for upper thoracic esophageal cancer .
4. Age ≧ 18 ys
5. KPS ≧ 60%
6. Hemogram : WBC ≧ 4000/mm3 or ANC ≧ 2000 /mm3 and Platelet ≧ 100,000/mm3 . Biochemistry : GOT/GPT ≦ 3.5 times , Cr ≦ 1.5 mg/dl and Bilirubin ≦ 2.0 mg/dl .

Exclusion Criteria:

1. Invasion to surrounding organ ( T4 disease ) .
2. Distant metastasis , except M1a disease .
3. Patients who refuse operation .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-08; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Clinical and pathological response rates | 2000~2004

SECONDARY OUTCOMES:
Progression free survival | 2000~2004
overall survival | 2000~2004
Toxicity | 2000~2004

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hsu, M.D.,Ph.D., Principal Investigator — Department of Oncology, National Taiwan University Hospital; Ann-Lii Cheng, M.D.,Ph.D, Study Chair — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, Nationa Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Guo JC, Huang TC, Lin CC, Hsieh MS, Chang CH, Huang PM, Lee JM, Hsu FM, Chia-Hsien Cheng J, Wang HP, Yeh KH, Cheng AL, Hsu CH. Postchemoradiotherapy Pathologic Stage Classified by the American Joint Committee on the Cancer Staging System Predicts Prognosis of Patients with Locally Advanced Esophageal Squamous Cell Carcinoma. J Thorac Oncol. 2015 Oct;10(10):1481-9. doi: 10.1097/JTO.0000000000000651. PMID 26313683